CLINICAL TRIAL: NCT00001211
Title: Clinical Study of Oral Endosseous Titanium Implants in Edentulous Subjects
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 860015; 86-D-0015
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Ectodermal Dysplasia; Jaw, Edentulous
Keywords: Ectodermal Dysplasia; Edentulous; Endosseous; Implants; Mandibular Atrophy; Oral; Titanium
MeSH Terms: conditions — Ectodermal Dysplasia; Jaw, Edentulous; Mouth, Edentulous

SUMMARY:
The amendment to Clinical Protocol 86-D-0015, clinical study of Oral Endosseous Titanium Implants in Edentulous subjects, and patients with Ectodermal Dysplasia is to allow the Investigators to determine: (1) If placement of Endosseous Titanium Implants in pre-adolescent patients (age 7 to 10) will influence the growth and development of the craniomandibular complex. (2) The final position of the implant, the ability to fabricate prosthesis. (3) Body image, diet and perceived ease of chewing selected foods.

Selection of patients for participation in the study will be based on the number of congenitally missing teeth associated with Ectodermal Dysplasia. At least 16 permanent teeth must be congenitally missing. A total of 30 patients will be included.

A consent to participate in this study will be obtained from each patient:

18 & older - consent signed by patient

13-17 years - consent signed by parent, assent signed by patient

7-10 years - consent by parent, assent signed by child if capable of understanding or note on chart describing procedure used to obtain the child's assent to the study

DETAILED DESCRIPTION:
The amendment to Clinical Protocol 86-D-0015, clinical study of Oral Endosseous Titanium Implants in Edentulous subjects, and patients with Ectodermal Dysplasia is to allow the Investigators to determine: (1) if placement of Endosseous Titanium Implants in pre-adolescent patients (age 7 to 10) will influence the growth and development of the craniomandibular complex. (2) The final position of the implant, the ability to fabricate prosthesis. (3) Body image, diet and perceived ease of chewing selected foods.

Selection of patients for participation in the study will be based on the number of congenitally missing teeth associated with Ectodermal Dysplasia. At least 16 permanent teeth must be congenitally missing. A total of 30 patients will be included.

A consent to participate in this study will be obtained from each patient:

18 & older - consent signed by patient

13-17 years - consent signed by parent, assent signed by patient

7-10 years - consent by parent, assent signed by child if capable of understanding or note on chart describing procedure used to obtain the child's assent to the study

ELIGIBILITY:
Individuals with a need for replacement maxillary and mandibular complete dentures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 1986-01; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Guckes AD, Smith DE, Swoope CC. Counseling and related factors influencing satisfaction with dentures. J Prosthet Dent. 1978 Mar;39(3):259-67. doi: 10.1016/s0022-3913(78)80092-4. No abstract available. PMID 273089
- [Background] Bolender CL, Swoope CC, Smith DE. The Cornell Medical Index as a prognostic aid for complete denture patients. J Prosthet Dent. 1969 Jul;22(1):20-9. doi: 10.1016/0022-3913(69)90268-6. No abstract available. PMID 5254404
- [Background] Bergman B, Carlsson GE. Review of 54 complete denture wearers. Patients' opinions 1 year after treatment. Acta Odontol Scand. 1972 Oct;30(4):399-414. doi: 10.3109/00016357209002493. No abstract available. PMID 4569753